CLINICAL TRIAL: NCT03249298
Title: Comparison of Crystaloids and Colloids for Fluid Optimization in Patients Undergoing Neurosurgical Procedure
Brief Title: Fluid Optimization With Crystalloids and Colloids in Neurosurgery
Acronym: KOKR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Jasmina Markovic Bozic, MD, PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OBKRGKOAIT216
Record Dates: First submitted 2017-04-07; First posted 2017-08-15 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — sterofundin; HES 130-0.4

STUDY DESIGN:
Intervention Model Description: one group will get crystalloids and one grou will get colloids for fluid optimisation

ARMS (2):
- Crystalloids (Active Comparator): Bolus of crystalloids
  Bolus of 250 ml crystaloids will be infused regarding the measures
  Interventions: Drug: Sterofundin (Bolus of crystalloids)
- Colloids (Active Comparator): Bolus of colloids
  Bolus of 250 ml colloids will be infused regarding the measures
  Interventions: Drug: Voluven (Bolus of colloids)

INTERVENTIONS:
Drug: Sterofundin (Bolus of crystalloids) — Bolus of 250 ml crystaloids infused regarding the measures
  Other Names: Sterofundin
  Arms: Crystalloids
Drug: Voluven (Bolus of colloids) — Bolus of 250 ml colloids infused regarding the measures
  Other Names: Voluven
  Arms: Colloids

SUMMARY:
Fluid optimization in neurosurgical patients has an important impact on preservation of cerebral perfusion pressure and minimization of cerebral oedema during and after the craniotomy. The investigators would like to know if crystalloids or colloids are equally useful for goal directed therapy in this patients. The investigators will record haemodynamic stability, volume loading and postoperative complications and compare two groups of patients. One group will be optimised with crystalloids and the second with colloids. The investigators will compare also hospital stay and mortality in the two groups.

DETAILED DESCRIPTION:
Hemodynamic stability and maintenance of cerebral perfusion pressure (CPP) are important in neurosurgical patients. Fluid management includes maintenance of intravascular volume, preservation of cerebral perfusion pressure and minimization of cerebral oedema. Fluid management of the neurosurgical patient has advanced from "run them dry" to "run them isovolaemic, isotonic and iso-oncotic, but the induction of potential complications by current strategies are still unknown. Advanced techniques provide goal directed fluid therapy which is currently the gold standard in fluid strategy. In patients undergoing craniotomy diuretics, preoperative fasting, induction of general anaesthesia and intraoperative bleeding may lead to hypovolemia and poor cerebral perfusion. On the other hand fluid overload increases complications and hospital stay after surgery. It is, therefore, important that optimal fluid levels are achieved.

The aim of the study was to compare intraoperative hemodynamic stability, volume loading and postoperative complications between group optimised with crystalloids and group optimised with colloids in patients undergoing neurosurgical procedure. The investigation will include 80 patients, 40 optimised with crystalloids and 40 with colloids.

Hemodynamic stability, volume loading, pooperative complications, hospital stay and mortality will be monitored during and aftre the surgery.

ELIGIBILITY:
Inclusion Criteria:

* neurosurgery (tumour, vascular, adenoma), haemodynamic stability

Exclusion Criteria:

* arrhythmia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Consumption of optimisation fluid | During surgery
  Investigators will record the number of interventions with fluid boluses and volume of optimisation fluid

SECONDARY OUTCOMES:
Postoperative complications | From the first day until 15 day after the surgery
  The investigators will record the incidence of postoperative complications Complications in different organs will be recorded (nevrological, pulmological, cardiovascular, haematological, infection, wound). The investigator will evaluate the days in the hospital after the surgery and the mortality rate (the number of deaths) for the 15 days after the surgery or until death or the dissmision.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No